CLINICAL TRIAL: NCT04496856
Title: The Effects of Whey Protein and Collagen on Fat Free Mass, Muscle Strength and Wound Healing in Elderly Patients Undergoing Elective Knee- or Hip Surgery
Brief Title: Effects of Whey and Collagen on FFM, Muscle Strength and Wound Healing in Elderly Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ValleKollagen
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hip Arthritis; Sarcopenia; Knee Arthritis
Keywords: Hip Arthroplasty; Collagen; Whey protein; Knee Arthroplasty
MeSH Terms: conditions — Sarcopenia | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen (Experimental): Participants of this arm are going to consume 30 g of collagen peptides daily for 30 days
  Interventions: Dietary Supplement: Whey protein and Collagen supplementation
- Whey Protein (Experimental): Participants of this arm are going to consume 30 g of whey protein daily for 30 days
  Interventions: Dietary Supplement: Whey protein and Collagen supplementation

INTERVENTIONS:
Dietary Supplement: Whey protein and Collagen supplementation — Participants of each arm will consume 30 g daily of the assigned protein supplementation for 30 days. The protein supplementation will be given as protein powder which the participants will have to dissolve in cold drinks. During the intervention fat free mass, muscle strength, functional ability, wound healing and life quality of the participants will be monitored.

SUMMARY:
The purpose of the study is to compare the effect of whey protein and collagen on fat free mass, muscle strength, functional ability, wound healing and life quality in elderly patients undergoing elective knee- or hip surgery (defined as elective knee- or hip arthroplasty). The patients are admitted at the department of Orthopaedic Surgery at Herlev Gentofte Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+ years
* Scheduled elective knee- or hip surgery
* Must be able to understand and speak danish
* Must be able to chew and swallow food with a regular consistency
* Must be able to consume the assigned protein supplementation
* Must be able to consent participation

Exclusion Criteria:

* Vegan
* Demensia
* Critical complications to the surgery which prevents the patient from participating in the rehabilitation program
* Plasma-creatinin above 250 micromol/L
* Palliative patients
* Known intolerance of whey protein and/or collagen
* Patients with a pacemaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The difference in fat free mass | Weekly for 30 days
  The outcome will be monitored through BIA and the development of fat free mass in the operated leg will be compared to the development of fat free mass in the non-operated leg.

SECONDARY OUTCOMES:
Wound healing | Weekly for 30 days
  The amount of days until the wound is healed (defined as: the epithelium is covered without crust). This will be monitored trough pictures and assessed on a scale from 1-5 by a masked doctor.
Redness and infection | Weekly for 30 days
  The redness and infection around the wound assessed on a scale from 1-5 by a masked doctor through pictures.
Handgrip strength | Weekly for 30 days
  Handgrip strength measured by a handdynanometer (SAEHAN) in kg and percentage
Extension strength of quadriceps femoris | Weekly for 30 days
  Measured in amounts of repetitions of 0.5 or 1.0 kg.
Life quality | Weekly for 30 days
  Measured trough EuroQol-5D-5L
Difference in functional ability (NMS) | Weekly 30 days
  Assessed by New mobility score
Difference in Chair stand test | Weekly for 30 days
  Measured by amount of repetitions

OTHER OUTCOMES:
Palatability of the protein supplementation | 30 days
  Assessed on a scale from 1-5
Consistency of the protein supplementation | 30 days
  Assessed on a scale from 1-5
Compliance of the protein supplementation intake | Weekly for 30 days
  Assessed trough a weekly form, which the participants will fill in
Rapported side effects | 30 days
  Participants will be informed to rapport if they experience any side effects throughout the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev/Gentofte Hospital, Gentofte Municipality, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided